CLINICAL TRIAL: NCT06647199
Title: Clinical Evaluation of Peri-Implant Tissues of CAD/CAM Milled PEEK, PMMA and Conventional Implant Assisted Overdentures
Brief Title: Evaluation of Peri-Implant Tissues of Different Implant Assisted Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Fatma Ahmad El Waseef, Associate professor of prosthodontics, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mansoura
Record Dates: First submitted 2024-10-15; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Peri-Implant Tissues

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAD/CAM Milled PEEK (Experimental): In the first group (CAD/CAM PEEK MODs), the mandibular master cast, mandibular trial denture, and maxillary denture were scanned using an intraoral digital scanner both separately while biting. The scanned data were saved in standard tessellation language (STL) file format and entered into the design software . The mandibular denture base and set-up were virtually designed. Based on the virtually created mandibular denture bases, the STL file of the designed denture base was imported into the milling machine to mill the prepolymerised PEEK discs to construct the CAD/CAM PEEK MOD base .
  Interventions: Procedure: the plaque index (PI); Procedure: the bleeding index (BI); Procedure: simpliﬁed gingival index(GI),
- CAD/CAM milled PMMA (Experimental): In the second group (CAD/CAM PMMA MODs), the STL file of the designed denture base was imported into the milling machine to mill the PMMA MOD base. The mandibular denture base and set-up were virtually designed. Based on the virtually created mandibular denture bases, the CAD/CAM PMMA MOD base was milled .Based on the scanned denture teeth, denture teeth were milled from tooth-coloured prepolymerized PMMA blocks, finished and polished, and then bonded with a methacrylate-based bonding agent into the PMMA milled base.
  Interventions: Procedure: the plaque index (PI); Procedure: the bleeding index (BI); Procedure: simpliﬁed gingival index(GI),
- conventional PMMA MOD (Experimental): the traditional heat-cured PMMA MOD was constructed. The waxed-up overdenture was processed in heat-cured PMMA resin using the compression mould technique.
  Interventions: Procedure: the plaque index (PI); Procedure: the bleeding index (BI); Procedure: simpliﬁed gingival index(GI),

INTERVENTIONS:
Procedure: the plaque index (PI) — Peri-implant soft tissue changes as regards plaque was assessed employing the modiﬁed plaque index (PI). Patients were evaluated clinically at the time of mandibular overdenture insertion (T0), 6 months (T1), 12 months (T2) and 3 years (T3) after denture insertion. Both plaque index (PI) and bleeding index (BI) were evaluated according to the Mombelli index , and gingival index (GI) according to the modified Silness and Loe index. Measurements were taken from the buccal, lingual, mesial, and distal aspects of each implant. All the clinical parameters were measured from the four aspects using a graduated periodontal probe (Hawe Perio-Probe, Kerr), and the sum total of the four readings was divided by four to obtain the mean value. The distance between the marginal border of the peri-implant mucosa and the tip of the probe was measured and considered as pocket depth (PD).
Procedure: the bleeding index (BI) — Peri-implant tissue changes as bleeding score was assessed employing the bleeding index (BI) . Patients were evaluated clinically at the time of mandibular overdenture insertion (T0), 6 months (T1), 12 months (T2) and 3 years (T3) after denture insertion. Both plaque index (PI) and bleeding index (BI) were evaluated according to the Mombelli index , and gingival index (GI) according to the modified Silness and Loe index. Measurements were taken from the buccal, lingual, mesial, and distal aspects of each implant. All the clinical parameters were measured from the four aspects using a graduated periodontal probe (Hawe Perio-Probe, Kerr), and the sum total of the four readings was divided by four to obtain the mean value. The distance between the marginal border of the peri-implant mucosa and the tip of the probe was measured and considered as pocket depth (PD).
Procedure: simpliﬁed gingival index(GI), — Peri-implant soft tissue changes as regards gingival scores was assessed simpliﬁed gingival index(GI). Patients were evaluated clinically at the time of mandibular overdenture insertion (T0), 6 months (T1), 12 months (T2) and 3 years (T3) after denture insertion. Both plaque index (PI) and bleeding index (BI) were evaluated according to the Mombelli index , and gingival index (GI) according to the modified Silness and Loe index. Measurements were taken from the buccal, lingual, mesial, and distal aspects of each implant. All the clinical parameters were measured from the four aspects using a graduated periodontal probe (Hawe Perio-Probe, Kerr), and the sum total of the four readings was divided by four to obtain the mean value. The distance between the marginal border of the peri-implant mucosa and the tip of the probe was measured and considered as pocket depth (PD

SUMMARY:
The researchers will perform a parallel randomized, clinical trial involving completely edentulous healthy patients. Each participant will receive four dental implants in the anterior mandible. According to the processing technique and denture base material, the patients will be classified into three groups. Group I: involves CAD/CAM milled poly ether ether ketone PEEK overdentures, Group II: involves CAD/CAM milled PMMA overdentures and Group III :involves conventional heat-cured poly methyl methacrylate PMMA overdentures. All assessments were carried out at delivery, 6 moths and one year after overdenture insertion to clinically evaluate the preiimplant tissues. .

DETAILED DESCRIPTION:
The study will be conducted to compare three different mandibular implant- assisted complete overdentures. These overdentures were constructed from three different materials and techniques: CAD/CAM-milled poly ether ether ketone (CAD/CAM PEEK MOD), CAD/CAM-milled poly methyl methacrylate (CAD/CAM PMMA MOD), and conventional heat-cured poly methyl methacrylate (conventional PMMA MOD) to clinically evaluate the preiimplant tissues.

The participants enrolled in the current study were randomly assigned to one of three groups based on the material and technique of their mandibular overdenture bases. All participants were delivered new sets of conventional complete dentures implied bilateral balanced occlusal scheme. They were well instructed to wear their dentures regularly for 3 months prior to implant installment ascribed to enhancement of the neuromuscular adaptation. For each patient, the mandibular denture was duplicated with clear auto- polymerizing acrylic resin to fabricate the mandibular surgical template with gutta percha markers. By employing CBCT, all patients were scanned conforming to the dual scan protocol .The implants were installed virtually parallel to each other and perpendicular to the occlusal plane at the areas of canines and lateral incisors .This was carried out using 3D image planning software . The surgical stent with four sleeves was constructed by rapid prototyping .It was placed over the proposed implant locations.Four dental implants were surgically placed in the anterior region of the mandible.Three months afterward, the mandibular impression was registered. The primary impression was recorded and poured to gain the primary cast. Upon that primary cast, a closed custom tray was constructed. The positioner attachments were screwed to the implants, the processing caps and metal housings were secured over them. The custom tray was border molded. By using silicon impression material , the deﬁnitive impression was made at the abutment level. The processing caps and the metal housings were removed from the impression which was being poured by extra hard scannable dental stone to obtain the master cast. Maxillomandibular relations were registered .This was accomplished with mandibular conventional record blocks opposed by the existing maxillary complete denture. Semi anatomical acrylic teeth were arranged employing bilateral balanced occlusion .The waxed overdentures were tried in the patient's mouth. According to the mandibular denture base material and processing technique of the prostheses, the subjects were divided into three groups: The first group (I) included 10 participants whose mandibular overdentures were fabricated by milling pre-polymerized poly ether ether ketone PEEK discs (CAD/CAM PEEK MODs, the second group(II) included 10 participants whose mandibular overdentures were constructed by milling prepolymerised PMMA resin discs (CAD/CAM PMMA MODs), while the third group(III) included 10 participants received conventionally constructed heat-cured poly methyl methacrylate mandibular PMMA overdentures (conventional PMMA MOD).All needed adjustments were executed at the insertion visit. This is to assure appropriate border extension, proper denture base ﬁt, even occlusal contact besides patient comfort. The female housing attachment was picked up to the ﬁtting surface of the mandibular overdenture bases using self-cure acrylic resin. The white processing cap was removed and replaced by a blue one. The mandibular overdentures were delivered to all participants according to their group.

Patients' evaluation Clinical evaluation Peri-implant soft tissue changes as regards plaque, bleeding, and gingival scores were assessed employing the modiﬁed plaque index (PI), bleeding index (BI) and simpliﬁed gingival index (GI), respectively. These indices were evaluated at prosthesis insertion (T0), 3 months (T1) , 6 months(T3) and 12 month (T4) after insertion. A calibrated pressure-sensitive plastic periodontal probe was utilized.

ELIGIBILITY:
Inclusion Criteria:

* Each selected subject fulfilled the following criteria:
* all subjects complained about insufficient retention and stability pertained to their mandibular dentures at their presentation;
* they had enough quantity and quality of bone in the mandibular lateral and canine areas to support the standard implants (14 mm in length and 3.6 mm in diameter) as verified by CBCT;
* they had healthy keratinized mucosa and a class I maxillomandibular relationship; besides, they had enough interarch space.

Exclusion Criteria:

* Diabetes, osteoporosis, and immunological deficiency
* subjects having head and neck radiation therapy or using anticoagulant medication.
* Those who had a history of temporomandibular joint dysfunction, which could interfere with appropriate function,
* those who smoked heavily were also excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Peri-Implant Tissues changes regarding plaque index (PI). | 2 years
  Peri-implant soft tissue changes as regards plaque was assessed employing the modiﬁed plaque index (PI).
Peri-Implant Tissues changes regarding The bleeding index (BI). | 2 years
  The bleeding index in accordance with Mombelli et al was used: score 0: no bleeding when using a periodontal probe; score1: isolated bleeding spots visible; score 2: a confluent red line of blood along the mucosal margin; score 3: heavy or profuse bleeding.
Peri-Implant Tissues changes regarding The gingival index (GI) | 2 years
  The modified Silness and Loe index, was used to calculate the gingival index:
  Score 0: normal peri implant mucosa; score 1: mild inflammation, slight color change, and slight edoema; score 2: moderate inflammation, redness, edoema, and glazing; and score 3: severe inflammation, marked redness and edoema, and ulceration.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Authors will share individual participant data if needed upon publishing process